CLINICAL TRIAL: NCT05305066
Title: Innovative Trial Designs, Multi-omics and Advanced Computational Prediction to Transform Clinical Care in RA
Brief Title: Stand UP to Rheumatoid Arthritis (SUPRA)
Acronym: SUPRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marie Hudson, MD (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Montreal General Hospital (Other); Lady Davis Institute (Other)
Responsible Party: Sponsor-Investigator, Marie Hudson, MD, Rheumatologist, Jewish General Hospital; Physician-scientist, Lady Davis Institute for Medical Research, Sir Mortimer B. Davis - Jewish General Hospital
Organization: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MP-05-2022-3107
Record Dates: First submitted 2022-02-26; First posted 2022-03-31 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Pragmatic trials; Feasibility
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept; Adalimumab; golimumab; Certolizumab Pegol; Interleukin-6 Inhibitors; tocilizumab; sarilumab; tofacitinib; upadacitinib; baricitinib

STUDY DESIGN:
Intervention Model Description: Two separate sub-studies will be conducted:
  Sub-study 1: Subjects who have failed conventional DMARDS will be randomised to receive therapy with TNFi or anti-IL6 using covariate adaptive randomization.
  Sub-study 2: Subjects who have failed TNFi will be randomised to receive therapy with anti-IL6 or JAKi using covariate adaptive randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sub-study 1 TNFi (Active Comparator): TNFi - any sub-cutaneous (sc) formulation, namely etanercept (receptor fusion protein), adalimumab (monoclonal antibody), golimumab (monoclonal antibody), or certolizumab (pegylated fragment of a monoclonal antibody)
  Interventions: Drug: TNFi
- Sub-study 1 Anti-IL6 (Active Comparator): Anti-IL6 receptor monoclonal antibodies - tocilizumab or sarilumab
  Interventions: Drug: Anti-IL6
- Sub-study 2 Anti-IL6 (Active Comparator): Anti-IL6 receptor monoclonal antibodies - tocilizumab or sarilumab
  Interventions: Drug: Anti-IL6
- Sub-study 2 JAKi (Active Comparator): JAKi - tofacitinib (JAK1/3 inhibitor), baricitinib (JAK 1/2 inhibitor) or upadacitinib (JAK1 inhibitor)
  Interventions: Drug: JAKi

INTERVENTIONS:
Drug: TNFi — TNFi - any sub-cutaneous (sc) formulation, namely etanercept (receptor fusion protein) 50 mg sc per week, adalimumab (monoclonal antibody) 40 mg sc every 2 weeks, golimumab (monoclonal antibody) 50 mg sc every month, or certolizumab (pegylated fragment of a monoclonal antibody) 400 mg sc at week 0, 2 and 4, and then 200 mg sc every 2 weeks or 400 mg sc every 4 weeks.
  Other Names: Etanercept; Adalimumab; Golimumab; Certolizumab
  Arms: Sub-study 1 TNFi
Drug: Anti-IL6 — Anti-IL6 receptor monoclonal antibodies - tocilizumab (if weight <100 kg: 162 mg SC every other week, followed by an increase to weekly based on clinical response; if weight ≥100 kg: 162 mg SC weekly) or sarilumab (200 mg SC once every 2 weeks)
  Other Names: Tocilizumab; Sarilumab
  Arms: Sub-study 1 Anti-IL6; Sub-study 2 Anti-IL6
Drug: JAKi — JAKi - tofacitinib (JAK1/3 inhibitor) 5 mg po bid, baricitinib 2 mg po qd (JAK 1/2 inhibitor) or upadacitinib 15 mg po qd (JAK1 inhibitor)
  Other Names: Tofacitinib; Upadacitinib; Baricitinib
  Arms: Sub-study 2 JAKi

SUMMARY:
Rheumatoid arthritis is a disabling arthritis that affects young women disproportionately. Although the physicians have some excellent treatments, they do not know which treatment is best for which patient. The investigators want to find ways to identify the right drug for the right patient at the right time. This is what personalized medicine is all about.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a complex, chronic disease of the immune system characterized by disfiguring and disabling arthritis. It affects predominantly women (3:1 ratio with men) and has its peak onset during their most productive years (ages 30-50). RA is associated with serious morbidity (including impaired fertility and pregnancy outcomes, disability, and depression) and premature mortality (particularly from cardiovascular and infectious causes). The Arthritis Alliance of Canada estimates that the cost of RA will exceed $30 billion in Canada in 2040.

First-line treatment of RA consists of conventional synthetic disease-modifying anti-rheumatic drugs (csDMARDs) with methotrexate considered as the gold standard. Yet, only 30% of patients will achieve adequate response to methotrexate and the majority will need additional treatment. The development of new biologic and targeted synthetic DMARDs (b/tsDMARDs) in the 20th century has transformed the treatment of RA. Anti-tumour necrosis factor (TNF)-α molecules were the first clinically successful biologic therapies for RA. Drugs targeting other signaling pathways (JAK-STAT, which work downstream of interferons), inflammatory cytokines (IL-6), as well as B cells and T cells have now also become available. Molecules with novel targets (eg. GM-CSF, CD40L) are in clinical trials.

Although hailed as 'game-changers' in patient care, the inconvenient truth is that even though nine different b/tsDMARDs are currently available to treat RA, 30% of patients will fail any particular drug. Moreover, physicians have no reliable way of predicting response and guiding treatment decisions. Clinical and genetic predictors have been the subject of intense research but these factors explain only a small portion of the observed variance in treatment response. Using the current trial-and-error approach, patients can cycle through multiple drugs before finally attaining disease control. This means months or years of suboptimal disease control and considerable losses in many domains including physical and emotional well-being, family and social networks, and occupational attainment. The lack of a personalized approach is particularly detrimental in RA because there is a narrow ''window of opportunity'' in the first 3-6 months of onset to control disease and optimize long term outcomes. In addition, failure to personalize treatment may also result in wasted spending on ineffective drugs, that cost up to $20,000 per patient per year, and exposing patients to unnecessary risks of adverse events, in particular serious infections.

There is a critical need to 1) transform the current 'trial-and-error' treatment paradigm, 2) explore novel predictors of b/tsDMARD response in RA and, 3) harness the power of advanced analytical strategies to personalize treatment decision-making and optimize outcomes in RA. The investigators propose a multi-pronged solution that combines innovative trial designs, multi-omics and advanced computational prediction to transform clinical care in RA.

The investigators propose to develop a new model of care and investigate new avenues, including sex and gender, diet, gut bacteria and environmental exposures, to make treatment decisions. The investigators will also use new methods of analyzing complex information. The highly talented research team has what is needed to transform the care of people living with RA.

In preparation for a full-scale study, the investigators propose this feasibility study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Arthritis that fulfills the 2010 ACR/EULAR classification criteria for RA;
* Failure to standard conventional synthetic DMARDs and eligible for second-line b/tsDMARDs (Sub-study 1) or failure to at least one TNF inhibitor and eligible for third-line b/tsDMARDs (Sub-study 2).

Exclusion Criteria:

* Prior b/tsDMARDs for Sub-study 1 or prior b/tsDMARDs other than TNF inhibitors for Sub-study 2;
* Contraindication to b/tsDMARD therapy, such as active infection or untreated latent TB, current malignancy, severe organ dysfunction, history of VTE (unless anticoagulated), high risk of cardiovascular disease, pregnancy/lactation;
* Overlap with another inflammatory disease requiring specific immunosuppressive therapy, such as lupus nephritis;
* Unable to provide consent or complete forms (alone or with assistance) in English or French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Rate of recruitment at two RA referral centers over 12 months | 12 months
  Feasibility outcome
Prompt access to drugs | 4 weeks
  Feasibility outcome
Proportion of participants adhering to the allocated treatment | 24 months
  Feasibility outcome
Proportion of eligible patients who are invited to participate by their physician | 12 months
  Physician acceptability outcome
Proportion of eligible patients who accept to participate | 12 months
  Patient acceptability outcome
Proportion of patients reaching SDAI <= 3.3 | 24 months
  Exploratory outcome
Proportion of patients reaching DAS28 LDA state | 24 months
  Exploratory outcome
Patient-reported outcomes (function, health-related quality of life, fatigue) | 24 months
  Exploratory outcome

CONTACTS AND LOCATIONS:
Overall Officials: Marie Hudson, MD, Principal Investigator — Sir Mortimer B. Davis - Jewish General Hospital
Locations (1):
- Sir Mortimer B. Davis Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Participants' study information and biological samples may be shared with researchers at this institution or other institutions for genetic, immunological, and other analyses (e.g. microbiome sequencing, biomarkers analyses, etc.).
Supporting Information: Study Protocol
Time Frame: After 2025, for 3 years
Access Criteria: The sharing of these samples will be done under specific research agreements; the samples and the data will be coded and confidentiality strictly protected.

REFERENCES:
- [Background] Loudon K, Treweek S, Sullivan F, Donnan P, Thorpe KE, Zwarenstein M. The PRECIS-2 tool: designing trials that are fit for purpose. BMJ. 2015 May 8;350:h2147. doi: 10.1136/bmj.h2147. No abstract available. PMID 25956159